CLINICAL TRIAL: NCT00822978
Title: A Double-Blind, Randomized, Placebo-controlled, Parallel-Group, Single and Multiple Dose-Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of ACHN-490 Injection Administered Intravenously in Healthy Volunteers
Brief Title: Phase 1 Study for Safety of ACHN-490
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Achaogen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: ACHN-490-001
Record Dates: First submitted 2009-01-13; First posted 2009-01-15 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: healthy; volunteers; subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACHN-490 Injection (Active Comparator): ACHN-490 Injection in escalating doses
  Interventions: Drug: ACHN-490 Injection vs placebo
- 2 (Placebo Comparator): Placebo is normal saline
  Interventions: Drug: ACHN-490 Injection vs placebo

INTERVENTIONS:
Drug: ACHN-490 Injection vs placebo — Escalating doses beginning with test dose given once, followed by 4 mg/kg with a single dose then multiple dose. Dose escalation to continue up to 15 mg/kg as long as the treatment is deemed safe.

SUMMARY:
This is a first-in-human phase 1 study to assess if ACHN-490 Injection is safe in people. Groups of people will receive either the study medication (ACHN-490) or a placebo (normal saline) as a single infusion. If the single dose is well tolerated then this group will receive 1 dose per day for up to 10 consecutive days. A new group of people will receive the study medication at a higher dose than the previous dose level as long as the previous dose was safe.

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* Within normal weight limits
* In good health with normal routine laboratory results
* Willing to not use media players (such as MP3 players) or devices with ear pieces and avoid exposure to loud noise

Exclusion Criteria:

* No ongoing medical conditions such as heart disease, high blood pressure, asthma, diabetes, seizures, or kidney problems
* No problems with hearing or balance
* No previous injury or surgery the the ears
* No family history of hearing loss before the age of 65
* Not taking any medication other than birth control medication
* Smokers or use of tobacco products
* Recent blood donor
* Allergy ot iodine, shellfish or aminoglycosides (a type of antibiotic)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2009-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Incident and severity of adverse events | 2 weeks after the last dose for each dose group

SECONDARY OUTCOMES:
Changes from baseline in kidney function, laboratory values, abd vital signs | single and multi-dose
Pharmacokinetic parameters | After single and multiple-dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Carter Brooks, MD, Principal Investigator — Jasper Clinic, Michigan
Locations (1):
- Jasper Clinic, Kalamazoo, Michigan, United States